CLINICAL TRIAL: NCT06337864
Title: Safety and Efficacy of Treatment With Large Neutral Amino Acids in Patients With Classical Phenylketonuria
Brief Title: Effect of Large Neutral Amino Acids in Adults With Classical Phenylketonuria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Prekulab Ltd ApS (Unknown)
Responsible Party: Principal Investigator, Allan Meldgaard Lund, Professor, MD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-24041030
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Brain Diseases; Brain Diseases, Metabolic; Brain Diseases, Metabolic, Inborn; Genetic Diseases, Inborn; Metabolism, Inborn Errors; Amino Acid Metabolism, Inborn Errors; Metabolic Disease; Phenylketonurias
MeSH Terms: conditions — Brain Diseases; Brain Diseases, Metabolic; Brain Diseases, Metabolic, Inborn; Genetic Diseases, Inborn; Metabolism, Inborn Errors; Amino Acid Metabolism, Inborn Errors; Metabolic Diseases; Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, crossover trial. Participants will be randomly assigned to receive either LNAA treatment or the classic dietary treatment for 8 weeks, followed by a washout period of 2 weeks before receiving the other intervention for 8 weeks. Additionally, a healthy control group will be recruited for baseline measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LNAA supplementation, Then Low-Phe diet (Experimental): Phase 1: LNAA Treatment Period (8 weeks) Each participant will be prescribed a specific dosage of LNAA tablets to be taken three times daily.
  Phase 2: Washout (2 weeks) Participants will follow a liberalized diet and refrain from taking any LNAA or amino acid supplement.
  Phase 3: Low-Phe diet (8 weeks) Each participant will follow a low-phenylalanine diet. LNAA therapy will not be administered during this phase.
  Interventions: Other: PreKUnil® LNAA Medical Food for PKU
- Low-Phe diet, Then LNAA supplementation (Experimental): Phase 1: Low-Phe diet (8 weeks) Each participant will follow a low-phenylalanine diet. LNAA therapy will not be administered during this phase.
  Phase 2: Washout (2 weeks) Participants will follow a liberalized diet and refrain from taking any LNAA or amino acid supplement.
  Phase 3: LNAA Treatment Period (8 weeks) Each participant will be prescribed a specific dosage of LNAA tablets to be taken three times daily.
  Interventions: Other: PreKUnil® LNAA Medical Food for PKU

INTERVENTIONS:
Other: PreKUnil® LNAA Medical Food for PKU — PreKUnil® LNAA Medical Food for PKU is a commercially available active LNAA treatment product for PKU.

SUMMARY:
The overall aim of this study is to evaluate LNAA treatment as a potential alternative to conventional dietary treatment for PKU. This study investigates the effects of LNAA treatment compared to the classic dietary treatment on cerebral dopamine synthesis in patients with classic PKU. We will assess LNAAs effectiveness on neurotransmitter synthesis, cognitive function, mental health, and safety, compared to the standard diet.

DETAILED DESCRIPTION:
Standard treatment for Phenylketonuria (PKU) involves a lifelong, phenylalanine-restricted diet. Strict adherence to the diet is crucial, but often challenging. Large neutral amino acid (LNAA) supplementation is a potential alternative therapeutic approach for PKU management. The proposed mechanism involves competitive inhibition of phenylalanine (Phe) transport across the blood-brain barrier by high-dose LNAA, leading to reduced brain Phe levels. However, further investigation is needed to validate its efficacy and safety for PKU management.

A randomized, open-label, crossover trial will be conducted to assess the safety and efficacy of LNAA supplementation in PKU patients. After completion of the crossover study, participants will have the option to participate in an open-label extension study aimed at evaluating the long-term safety and efficacy of LNAA.

A healthy control group will be recruited to obtain baseline outcome measures. This project is expected to provide much-needed insights into the potential of LNAA in PKU management. The study also aims to gain a deeper understanding of the underlying pathophysiology of the disease. Finally, this work could lead to more personalized management strategies for PKU patients.

ELIGIBILITY:
Patients ≥ 18 years of age with Classical PKU molecularly confirmed via the finding of two pathogenic variants in the phenylalanine hydroxylase (PAH) gene and/or historical evidence of Phe concentrations ≥1200 μmol/L in the medical history

Inclusion Criteria:

* Treatment initiation within the first month of life
* Intelligence quotient over 84, based upon the baseline neuropsychological evaluation
* Conventional dietary treatment up to minimum 15 years of age
* Signed informed consent
* Willing and able to comply with the protocol and study procedures

Exclusion Criteria:

* Unable or unwilling to adhere to the requirements of the study
* A female who is pregnant or breastfeeding or planning to get pregnant during the study period
* Concomitant medication that may interfere with the PET analysis, as judged by the investigator
* A serious neuropsychiatric disease that could interfere with the subject's ability to participate in the study at the discretion of the investigator
* Concomitant treatment with BH4 supplementation (sapropterin) or Pegvaliase-pqpz (PALYNZIQ)
* Failing to submit at least one blood Phe home sample during the year before study initiation
* Standard MRI contraindications
* Body weight over 110 kg

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic positron emission tomography (PET) imaging with the fluorine-18-labeled tracer [18F]-(E)-N-(3-iodoprop-2-enyl)-2β-carbofluoroethoxy-3β-(4'-methyl phenyl)nortropane ([18F]FE-PE2I) | Crossover study: at 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Change in specific binding ratio of dopamine transporter (DaT) with [18F]FE-PE2I

SECONDARY OUTCOMES:
Urine peripheral biomarkers of neurotransmitters | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  6-sulfatoxymelatonin and dopamine
Incidence and severity of treatment-emergent adverse events (TEAEs) | Baseline to week 80
  Subjects with at least one TEAE or serious TEAE
Adult attention deficit hyperactivity disorder (ADHD) Self-Report Scale (ASRS v1.1) | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Patient-Reported Outcome Measure of attention in adults, 0-23, lowest is best
Symptom Checklist-90-Revised (SCL-90-R) | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Patient-Reported Outcome Measure of psychopathological symptoms, percentile, lowest is best
Neuropsychological testing of flexibility and verbal fluency | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Change in flexibility and verbal fluency using the Delis-Kaplan Executive Function System (D-KEFS) customized for study
Behaviour Rating Inventory of Executive Function - Adult version (BRIEF-A) | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Patient-Reported Outcome Measure of executive functioning (ages 18 to 90), percentile, lowest is best
PKU-QOL Questionnaire Adult version | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Patient-Reported Outcome Measure of the impact of PKU and the PKU diet on quality of life
Computerized neuropsychological testing (responses over study iPad) | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Cambridge Neuropsychological Test Automated Assessment Battery (CANTAB) customized for study

OTHER OUTCOMES:
Brain Magnetic Resonance Imaging (MRI) | Inclusion
  Percent of patients with anatomic anomalies on MRI of the brain
Wechsler Adult Intelligence Scale (WAIS) - IV | Inclusion
  Baseline measure of cognitive ability, 40-160, highest is best
Fasting plasma amino acids, dried blood spots (finger-prick method) | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Biomarkers such as the plasma Phe, Phe/Tyr ratio, Tyr/LNAA, Trp/LNAA ratio
Adherence to dietary treatment | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  3-day diet record
Brain perfusion measures | Crossover study: at baseline, 8, 10 and 18 weeks from baseline, Extension study: at 12 months from baseline
  Dynamic PET Imaging differences between groups and with intervention

CONTACTS AND LOCATIONS:
Overall Officials: Allan Lund, Professor, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Center for Inherited Metabolic Diseases, Copenhagen
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No